

# **Non-interventional Study Protocol**

| <b>Document Number:</b> | c10705101-01 |
|---|---|
| BI Study Number: | 1237.58 |
| BI Investigational Product(s): | Spiolto <sup>®</sup> Respimat <sup>®</sup> |
| Title: | Assessment of physical functioning and handling of Spiolto <sup>®</sup> Respirat <sup>®</sup> in patients with chronic obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine clinical practice. |
| Brief lay title | OTIVACTO NIS SPAIN |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | 13 June 2016 |
| PASS: | No |
| EU PAS register | Not yet available |
| number: | (study will be registered in EU PAS Register (ENCePP) and clinicaltrials.gov) |
| Active substance: | R03AL06 |
| | Tiotropium bromide + Olodaterol |
| Medicinal product: | Spiolto® Respimat® 2.5 microgram/2.5 microgram, inhalation solution; tiotropium/olodaterol |
| Product reference: | NL/H/3157/001/DC |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | MAH: Boehringer Ingelheim International GmbH Binger Straße 173 55216 Ingelheim am Rhein |
| | This study is initiated, managed and sponsored by: |
| | Boehringer Ingelheim España, S.A<br>C/ Prat de la Riba, 50<br>08174 Sant Cugat del Vallés (Barcelona) |
| Joint PASS: | No |
| Research question and | Primary objective |
| objectives: | The objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto® |

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | Respimat® after approximately 6 weeks. |
|---|---|
| | Secondary objectives |
| | A secondary objective is to evaluate the patient's general condition (physician's evaluation) at visit 1 (baseline visit at the start of the study) and at visit 2 (final visit approx. 6 weeks after visit 1), as well as patient satisfaction with Spiolto® Respimat® at visit 2. |
| Country of study: | Spain |
| Author: | (Outsourced Trial Clinical Monitor) |
| | Mobile: |
| Marketing authorisation holder(s): | Boehringer Ingelheim International GmbH Binger Str. 173 D-55216 Ingelheim am Rhein Germany |
| MAH contact person in | Not applicable |
| case of PASS: | Not applicable |
| EU-QPPV in case of PASS: | Not applicable |
| Signature of EU-QPPV in case of PASS: | Not applicable |
| Date: | 13 June 2016 |
| Page 2 of 42 | |
| Proprietary confidential information | |

© 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| 1. | TABL | E OF CONTENTS | 3 |
|------|--------|----------------------------------|----|
| 2. | LIST ( | OF ABBREVIATIONS | 5 |
| 3. | RESPO | ONSIBLE PARTIES | 6 |
| 4. | ABST | RACT | 7 |
| 5. | AMEN | NDMENTS AND UPDATES | 10 |
| 6. | MILES | STONES | 11 |
| 7. | RATIO | ONALE AND BACKGROUND | 12 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES | 14 |
| 9. | RESEA | ARCH METHODS | 15 |
| 9.1 | STU | JDY DESIGN | 15 |
| 9.2 | SET | TTING | 15 |
| 9 | .2.1 | Study sites | 15 |
| 9 | .2.2 | Study population | 15 |
| 9 | .2.3 | Study visits | 16 |
| 9 | .2.4 | Study discontinuation | 17 |
| 9.3 | VA | RIABLES | 17 |
| 9 | .3.1 | Exposures | 17 |
| 9 | .3.2 | Outcomes | 18 |
| 9 | .3.2.1 | Primary outcomes | 18 |
| 9 | .3.2.2 | Secondary outcomes | 18 |
| 9 | .3.3 | Covariates | 19 |
| 9.4 | DA | TA SOURCES | 19 |
| 9.5 | STU | JDY SIZE | 19 |
| 9.6 | DA | TA MANAGEMENT | 20 |
| 9.7 | DA | TA ANALYSIS | 20 |
| 9 | .7.1 | Main analysis | 20 |
| 9.8 | QU | ALITY CONTROL | 22 |
| 9.9 | LIN | ITATIONS OF THE RESEARCH METHODS | 22 |
| 9.10 | OT | HER ASPECTS | 23 |
| 9 | 10.1 | Data quality assurance | 23 |

# **Non-interventional Study Protocol**

#### BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies 9 10 2 Study records 23 9.10.2.1 Source documents 23 9.10.2.2 9.10.3 10.1 10.2 MANAGEMENT AND REPORTING OF ADVERSE EVENTS & ADVERSE 11. 11.1 11.2 11.3 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS 12. 31 REFERENCES 32 13. PUBLISHED REFERENCES. 32 13.1 13.2 

#### **Non-interventional Study Protocol**

#### BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special Interest

CML Local Clinical Monitor

COPD Chronic Obstructive Pulmonary Disease

CRA Clinical Research Associate eCRF Electronic Case Report Form DMP Data Management Plan

EU European Union

FDC Fix Dose Combination

FEV<sub>1</sub> Forced expiratory volume in one second

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice

GOLD Global Initiative for Chronic Obstructive Lung Disease

ICH International Conference on Harmonisation

ICS Inhalative Corticosteroids
IEC Independent Ethics Committee

ISF Investigator Site File

LABA Long-acting beta<sub>2</sub> adrenoceptor agonist LAMA Long-acting muscarinic antagonist

MedDRA Medical Dictionary for Drug Regulatory Activities

mMRC Modified Medical Research Council Scale

NIS Non-Interventional Study

PF-10 Physical Functioning patient questionnaire

PGE Physician's Global Evaluation

SAE Serious Adverse Event SAP Statistical Analysis Plan

SF-36 36-Item Short Form Health Survey SGRQ St George's Respiratory Questionnaire SmPC Summary of Product Characteristics

TDI Transition Dyspnea Index WHO World Health Organisation

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. RESPONSIBLE PARTIES

| Therapeutic Area Respiratory Medicine (TA) | |
|---|---|
| Team Member Medical Affairs (TM MA) | |
| Team Member Epidemiology (TM Epi) | _ |
| Global Epidemiology ( GEpi) | |
| Therapeutic Area Risk Management (TA RM), and Pharmacovigilance Working Group (PVWG) chairperson | _ |
| GPV Study Coordination | _ |
| Trial Statistician (TSTAT) | · |
| Trial Data Manager (TDM) | · |
| Trial Programming | · |
| Team Member Medicine (TMM) | - |
| Trial Clinical Monitor (TCM) | (outsourced) |
| Coordinating Investigators (CI) in Spain | |

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of company | • | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Spiolto® Respimat® | | | |
| Name of active ing<br>Tiotropium bromid<br>Olodaterol (BI 174 | e (Ba679) + | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 13 Jun 2016 | 1237.58 | 1.0 | Not applicable |
| Title of study: | in patients with ch | vsical functioning and handli<br>ronic obstructive pulmonary<br>ronchodilation in routine clin | disease (COPD) requiring |
| Rationale and background: | Reduced physical activity resulting in deconditioning and restricted physical functioning is a common constraint of patients with moderate to very severe COPD. Clinical studies investigating treatment with Spiolto <sup>®</sup> Respimat <sup>®</sup> and its single components have shown significant improvements in exercise capacity in patients with COPD. Real-world data on the effects of a fixed-dose combination (LABA+LAMA) therapy with tiotropium and olodaterol administered in a single device, in COPD patients who need treatment with two longacting bronchodilators, is not available. | | |
| Research question and objectives: | The primary objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto <sup>®</sup> Respimat <sup>®</sup> after approximately 6 weeks. | | |
| | A secondary objective is to evaluate the patient's general condition (physician's evaluation) at visit 1 (baseline visit at the start of the study) and at visit 2 (final visit approx. 6 weeks after visit 1), as well as patient satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> at visit 2. | | |
| Study design: | Open-label observational study, including COPD patients in Spain receiving treatment with Spiolto <sup>®</sup> Respimat <sup>®</sup> for approximately 6 weeks, which is the average time between two medical consultations. | | |
| Population: | COPD patients requiring a fixed combination therapy of two long-acting bronchodilators (LAMA + LABA) according to approved SmPC and GOLD guidelines. | | |
| Variables: | <ul> <li>Patient demographics (age, gender, height &amp; weight)</li> <li>Concomitant diseases / Comorbidities</li> <li>Concomitant medication</li> <li>General condition of patient based on Physician's Global Evaluation (PGE)</li> </ul> | | |

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of company: Boehringer Ingelheim | | | |
|---|---|---|---|
| Name of finished medicinal product: Spiolto® Respimat® | | | |
| Name of active ingredient:<br>Tiotropium bromide (Ba679) +<br>Olodaterol (BI 1744) | | | |
| Protocol date: Study number: | | Version/Revision: | Version/Revision date: |
| 13 Jun 2016 1237.58 | | 1.0 | Not applicable |
| | <ul> <li>Smoking history</li> <li>Exacerbations</li> <li>Breathlessness based on mMRC score</li> <li>Physical Functioning based on PF-10 scores</li> <li>Patient satisfaction with Spiolto® Respimat®</li> <li>Safety; ADR (serious and non-serious), fatal AEs, pregnancies</li> <li>GOLD spirometric classifications (1, 2, 3, 4)</li> <li>GOLD patient groups (A, B, C, D)</li> </ul> | | |

# Non-interventional Study Protocol

BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of compan | y: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Spiolto® Respimat® | | | |
| Name of active in<br>Tiotropium bromic<br>Olodaterol (BI 174 | de (Ba679) + | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 13 Jun 2016 | 1237.58 | 1.0 | Not applicable |
| Data sources: Study size: | To be completed by the physician: Patient demographics Patient medical files Physician's Global Evaluation (PGE) at visit 1 and visit 2 To be completed by the patient at Visit 1: mMRC breathlessness scale To be completed by the patient at visit 2 only: Patient satisfaction survey To be completed by the patient at visit 1 and at visit 2: Physical Functioning Questionnaire (PF-10) It is planned that data of approximately 1000 patients from | | |
| Data analysis: | approximately 200 sites (primary care) in Spain will be collected. Primary outcomes: "Therapeutic success" at visit 2 (10-point increase in the PF-10 score between visit 1 and visit 2). Secondary outcomes: - Changes in the PF-10 score from visit 1 to visit 2 - General condition of the patient, evaluated by the physician (PGE - score) at visit 1 and visit 2. - Patient satisfaction with Spiolto® Respimat® at visit 2. | | |
| Milestones: | Planned end of dat | nta collection: October-2016<br>ta collection: July-2017<br>y report: November-2017 | |

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. AMENDMENTS AND UPDATES

None

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------|---------------|
| Start of data collection | October 2016 |
| End of data collection | July 2017 |
| Final report of study results: | November 2017 |

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

COPD is defined as a preventable and treatable disease of the airways, with significant systemic consequences. Inactivity is believed to be crucial to the development of the extrapulmonary effects of the disease like skeletal muscle weakness, osteoporosis and cardiovascular disease. Recent data suggest that patients suffering from COPD with low levels of physical activity have increased risk for hospital admission and have significantly enhanced mortality. Epidemiological data suggest that this may directly or indirectly lead to more rapid decline in lung function [R13-3633].

Physical activity is reduced early in the disease progression, as of GOLD Stage 2 [R13-3633]. More recent evidence from large placebo controlled clinical trials indicates that COPD patients are experiencing a steeper absolute decline in lung function with GOLD 2 airflow limitation than with GOLD 3 and 4 [R15-5015]. All these observations suggest the importance of early optimal treatment of the disease.

Long-acting bronchodilators, such as long-acting muscarinic antagonists (LAMAs), are the cornerstone of maintenance therapy for patients with moderate to very severe chronic obstructive pulmonary disease (COPD) whose symptoms are not adequately controlled by short-acting bronchodilators alone [P13-05794, P14-01052].

An option recommended by GOLD guideline for patients not adequately controlled on a single long-acting bronchodilator is to combine a LAMA with a long-acting  $\beta$ 2-agonist (LABA) [P14-01052]. This has prompted the development of combining LAMA+LABA as fixed-dose combinations [P13-05794]. The rationale for combining bronchodilators with different mechanisms is based on the notion of additive relaxation of airway smooth muscle by direct inhibition of cholinergic activity and functional antagonism of bronchoconstriction through  $\beta$ 2-adrenergic pathways, with the expectation of an increase in the degree of bronchodilation for equivalent or lesser side effects. Several recent studies have provided evidence in support of this increased bronchodilatory effect when LABAs are added to LAMAs.

When long acting beta-agonists (LABA) and long acting muscarinic antagonists (LAMA) with similar or equivalent posologies are combined, the opportunity exists for offering a simpler and more convenient administration regimen with the development of fixed combinations within the same inhaler device. Fixed-dose combinations of a short-acting  $\beta$ 2–agonist and a short-acting anticholinergic have been developed and have been shown to be safe, efficacious and convenient for the patient (e.g., Berodual®: Fenoterolhydrobromid + Ipratropiumbromid, Combivent®: salbutamol + ipratropium bromide; [P94-1346]). Olodaterol is a highly selective and nearly full  $\beta$ 2 agonist [P10-07776, P11-07720] that provides 24-h bronchodilation in patients with COPD [P13-11467, P13-14112, P13-11346, P13-11345]. Olodaterol is also associated with symptomatic benefit [P13-11341] and enhanced exercise capacity [P13-14109].

The complementary modes of action of tiotropium and olodaterol have previously been demonstrated in animal models, phase II clinical trials and during the Phase IIIa programs [P10-09337, P14-12073, P10-14042, P13-02357].

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In the Phase III program the additional benefits of the tiotropium + olodaterol fixed-dose combination (FDC) over its mono-components has been assessed on lung function, quality of life (St. George's Respiratory Questionnaire -SGRQ), dyspnea (Transition Dyspnea Index-TDI) and exercise endurance time. Another clinically important potential benefit of the tiotropium + olodaterol FDC over the mono components, the impact on exacerbations of COPD, is currently evaluated in a Phase IIIb trial.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8. RESEARCH QUESTION AND OBJECTIVES

The contribution of physical inactivity to disability in COPD is difficult to distinguish from disease progression; however, it is clear that physical activity is significantly lower in patients with COPD than in healthy controls [R13-3633].

COPD prevents patients from carrying out daily activities due to exercise intolerance, which is often attributed to limited pulmonary ventilation. Physical inactivity may be related to avoidance of exertion as a result of fear of dyspnea. Furthermore, physical inactivity has been associated with skeletal muscle weakness and exercise intolerance [R15-4559, R15-4561].

The loss of physical activity in COPD is also associated with increased mortality. Data from a study of 2386 patients with COPD demonstrated that, following adjustment for relevant confounders, subjects who reported low, moderate or high physical activity had a significantly lower risk of all-cause mortality than those with very low physical activity (p = 0.001) [R15-4564]. Clinical studies of both Spiriva® [P13-04267, P05-09483, P13-14109] and Striverdi® Respimat® in COPD patients have demonstrated significant improvement in exercise capacity [P13-14109].

The benefits of tiotropium + olodaterol FDC have been studied in controlled Phase III programs on exercise endurance, however, data regarding physical activity when treated with Spiolto<sup>®</sup> Respirat<sup>®</sup> is not available from a real world setting.

The primary objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto<sup>®</sup> Respirat<sup>®</sup> after approximately 6 weeks in routine clinical practice.

The secondary objectives are to evaluate the patient's general condition (physician's evaluation) at visit 1 (baseline visit at the start of the study) and at visit 2 (final visit approx. 6 weeks after visit 1), as well as patient satisfaction with Spiolto<sup>®</sup> Respirat<sup>®</sup> at visit 2.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is an observational study as the medicinal product is prescribed according the normal clinical practice. The patient's assignment to a particular therapeutic strategy is not decided in advance by the study protocol but it will be determined by routine clinical practice and the decision to prescribe a particular medicinal product will be clearly dissociated from the decision to include the patient in the study. No other clinical intervention (diagnostic or clinical follow up) than the usual clinical practice will be applicable in the study.

This is a self-controlled study design enrolling consented COPD patients who will be treated with Spiolto<sup>®</sup> Respirat<sup>®</sup> according to the approved SmPC.

Patients will be enrolled consecutively and will be followed over an observational period of approx. 6 weeks.

Every physician is invited to enroll the first consecutive patients he/she chooses to treat with Spiolto® Respimat®. The decision to treat will be taken independently of participation in this NIS and will be made before participation is considered.

#### 9.2 SETTING

#### 9.2.1 Study sites

It is planned that data of approximately 1.000 patients from approximately 200 sites (primary care sites) in Spain will be collected. Site selection will be performed to reflect routine COPD care in order to secure representativeness of the COPD population. The inclusion of five patients is planned per investigator.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the Investigator Site File (ISF) irrespective of whether they have been treated or not.

#### 9.2.2 Study population

Patients can be included if all of the following criteria are met:

#### **Inclusion criteria**

- 1. Written informed consent prior to participation
- 2. Female and male patients  $\geq 40$  years of age
- 3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation (LAMA + LABA) treatment according to approved Spiolto<sup>®</sup> Respimat<sup>®</sup> SmPC and COPD GOLD guideline recommendation

#### **Exclusion criteria**

- 1. Patients with contraindications according to Spiolto<sup>®</sup> Respirat<sup>®</sup> SmPC
- 2. Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months

# Non-interventional Study Protocol

#### BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 3. Patients continuing LABA-iCS treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists
- 4. Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks
- 5. Pregnancy and lactation
- 6. Patients currently listed for lung transplantation
- 7. Current participation in any clinical trial or any other non-interventional study of a drug or device

#### 9.2.3 Study visits

Table 9.2.3:1: Visit flow chart and data collection parameters

| Parameter | Visit 1;<br>baseline<br>visit | Visit 2;<br>approx. 6<br>weeks after<br>baseline visit |
|---|---|---|
| Informed Consent | X | |
| Inclusion / Exclusion Criteria | X | |
| Patient demographics (age, gender, height, and weight) | X | |
| Start of COPD | X | |
| Number of exacerbations in the last 12 months | X | |
| Number of exacerbations leading to hospitalization in the last 12 months | X | |
| mMRC breathlessness scale | X | |
| Past COPD therapies (6 months before visit 1) | X | |
| Respimat® training (yes/no) | X | |
| COPD severity based on GOLD assessment <sup>1</sup> | X | |
| Smoking status | X | X |
| Concomitant diseases / Comorbidities | X | X |
| COPD related and other relevant concomitant medication | X | X |
| Physical functioning (PF-10) questionnaire, completed by patient | X | X |
| General condition of patient evaluated by Physician's Global Evaluation (PGE) | X | X |
| Safety: Adverse Drug Reactions (serious and non-serious), fatal AE, pregnancy | X | X |
| Patient satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> , survey completed by the patient | | X |
| Rational for Spiolto® Respimat® treatment discontinuation (if applicable) | | X |
| Continuation or discontinuation of treatment with Spiolto® Respimat® after the study (yes/no) | | X |

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

1 GOLD patient group (A, B, C or D) will be automatically calculated within the eCRF based on available exacerbation history, mMRC, and GOLD spirometric classification of airflow limitation based on post-bronchodilator FEV1 if available.

Baseline characteristics of patients being eligible and who gave Informed Consent, but were not treated in the study will also be collected.

#### 9.2.4 Study discontinuation

Boehringer Ingelheim reserves the right to discontinue the study or to remove a patient at a particular study site for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site.
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the study, or any other administrative reasons, i.e. lack of recruitment.
- 3. Violation of the protocol, the contract, or applicable laws and regulations for non-interventional studies, which could disturb the appropriate conduct of the NIS.

The investigator / the study site will be reimbursed for reasonable expenses incurred in case of study termination (except in case of the third reason).

#### 9.3 VARIABLES

### 9.3.1 Exposures

Tiotropium + olodaterol FDC is an aqueous solution of tiotropium and olodaterol contained in a cartridge. It is administered by using the Respimat® inhaler. One cartridge is used per inhaler, which is inserted into the device prior to first use. In pivotal clinical trials and for the intended marketed product, the clinical dose consists of two puffs once daily. The Respimat® inhaler uses mechanical energy to create a soft mist which is released over a period of approximately 1.5 seconds.

Tiotropium + olodaterol FDC was shown to be safe and well tolerated over 1 year in a moderate to very severe COPD population. The overall incidences of adverse events (AEs), serious adverse event (SAEs), fatal AEs, frequencies for cardiac events and major adverse cardiovascular event in the tiotropium + olodaterol FDC treatment group were similar to the mono-components. The nature and frequency of AEs in general was consistent with the disease under study. There were no results in the clinical development program suggesting the need for absolute contraindications for the combination product [P15-03349].

In conclusion, the clinical trials conducted to date have shown tiotropium + olodaterol FDC to be a safe, well tolerated and efficacious combination therapy according to treatment guidelines in a moderate to very severe COPD patient population [P15-04531, P15-03349]. The observed incremental bronchodilator response for the combination compared to the individual components translated into benefits that were meaningful to the patient, with improvements in several patient centered outcomes. For further information please refer to the SmPC of Spiolto® Respimat®.

# **Non-interventional Study Protocol**

#### BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.2 Outcomes

#### 9.3.2.1 **Primary outcomes**

"Therapeutic success" at visit 2 (10-point increase in the PF-10 score between visit 1 and visit 2).

#### 9.3.2.2 **Secondary outcomes**

- Changes in the PF-10 score from visit 1 to visit 2
- General condition of the patient, evaluated by the physician (PGE score) at visit 1 and visit 2.
- Patient satisfaction with Spiolto<sup>®</sup> Respirat<sup>®</sup> at visit 2.

The following parameters will be collected and assessed at visit 1 and/or visit 2:

- Patient demographics (age, gender, height & weight),
- Smoking status (current smokers, former smokers, and never smokers) and pack-years,
- Concomitant diseases / Comorbidities such as cardiovascular disease, diabetes mellitus, musculoskeletal impairment. renal diseases. liver diseases. osteoporosis. gastroesophageal reflux (GERD), or lung cancer,
- COPD related and other relevant concomitant medication such as beta-blockers, betaagonists, corticosteroids, or proton pump inhibitors,
- Reported exacerbations based on medical history in the last 12 months and exacerbations leading to hospitalization in the last 12 months,
- Assessment of the severity of breathlessness based on the Modified Medical Research Council Questionnaire (mMRC),
- Physical Functioning based on PF-10 scores\*, Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> to assess the overall satisfaction with Spiolto<sup>®</sup> Respirat<sup>®</sup> as well as specific inhalation from the device and device handling,
- General condition of patient based on Physician's Global Evaluation (PGE) to assess the general condition of the patient at the beginning and at the end of the study,
- Safety Reporting; Adverse Drug Reactions (serious and non-serious), fatal AEs, and pregnancies at the beginning and at the end of the study, as well as,
- GOLD spirometric classifications (1, 2, 3, 4) and GOLD patient groups (A, B, C, D) based on GOLD guidelines

\*The PF-10 is a sub-domain of the SF-36 and consists of 10 questions evaluating the extent of experienced restrictions while conducting usual activities. Each question of the PF-10 can be answered with "yes, limited a lot", "yes, limited a little", or "No, not limited at all", with a score of 1, 2, or 3. The scores over the 10 questions will be summed, resulting in a value between 10 (a patient answering all questions with "yes, limited a lot") and 30 (a patient answering all questions with "No, not limited at all"). The final sum of the individual scores will be standardized to a range of 0 to 100 using the following formula: 100\*(sum-10)/20.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.3 Covariates

Not applicable

#### 9.4 DATA SOURCES

Medical records collected through routine clinical care will be used to assess the inclusion/exclusion criteria of patients. Such medical records will be used for patient demographics, smoking history, collection of previous COPD medication, concomitant diseases, and concomitant medication.

All patients will be enrolled consecutively.

The treating physician will use the Physician's Global Evaluation (PGE) to evaluate the general condition of the patient on an 8-point ordinal scale from 1 (very poor) to 8 (excellent). PGE will be completed before and approx. 6 weeks after treatment initiation.

The modified Medical Research Council (mMRC) scale will be used to assess the breathlessness state of the patient before and after the treatment. The mMRC stage (0 to 4) collected from the patient, as well as the exacerbation history and the post-bronchodilator FEV<sub>1</sub>, will be used to automatically calculate the GOLD patient group (A, B, C, or D) in the eCRF.

The physical functioning (PF-10) questionnaire is a subscale of the validated 36-Item Short Form Health Survey and contains 10 questions about everyday physical activity and functioning. Patients will be asked to complete the PF-10, in order to evaluate their physical functioning before and after treatment with Spiolto<sup>®</sup> Respimat<sup>®</sup>.

A patient satisfaction survey will also be completed at visit 2, using a 7-point ordinal scale with divisions from very satisfied to very dissatisfied.

#### 9.5 STUDY SIZE

In a previous study, 205.426 (clinicaltrials.gov NCT 00699699): "Assessment of Physical Activity (PF10 Sub Domain of SF-36 Activity Score) and Tolerability in COPD Patients During Treatment With Spiriva® Respimat®), with over 1000 patients treated with Spiriva® Respimat®, therapeutic success (i.e., 10-point increase in the PF-10 score between visit 1 and visit 2) was achieved in 61% of the patients.

In this study, a lower therapeutic success rate is expected as patients may be already on maintenance treatment at baseline. Assuming a 50% therapeutic success rate and 900 patients, the 95% confidence interval for the therapeutic success rate would be between 46.7% (lower limit) and 53.3% (upper limit) (level of accuracy of  $\pm$  3.3%), basing the calculations on a binomial distribution.

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

To account for a 10% drop-out rate, the sample size is adjusted to 1.000 patients.

Calculations were performed with the PASS software package, version 2011.

#### 9.6 DATA MANAGEMENT

A data management plan (DMP) will be created to describe all functions, processes, and specifications for data collection, cleaning and validation. The electronic Case Report Forms (eCRFs) will include programmable edits to obtain immediate feedback if data are missing (also negative answers, unknown), out of range, illogical or potentially erroneous. These rules may encompass simple checks such as range validation or presence/absence of data. Concurrent manual data review may be performed based on parameters dictated by the DMP. Ad hoc queries to the sites may be generated and followed up for resolution. A source data quality audit may be initiated to ensure that the data in the database is accurate.

The database will be housed in a physically and logically secure computer system maintained in accordance with a written security policy. The system will meet the standards of the International Committee on Harmonization guideline E6R1 regarding electronic study data handling. Patient confidentiality will be strictly maintained.

#### 9.7 DATA ANALYSIS

#### 9.7.1 Main analysis

In this non-interventional study, cross-sectional data at study baseline and longitudinal follow-up data over 6 weeks will be collected for patients with chronic obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine clinical practice.

Baseline data will be described using a cross-sectional approach. Data from the longitudinal follow-up will be summarized descriptively. Due to the nature of this non-interventional study, there is no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses are descriptive in nature and confidence intervals and p-values from statistical models are used for exploratory purposes. No adjustments for multiple testing are made in the evaluation of statistical significance. Consequently, significant differences may be observed by chance alone and p-values should be interpreted as exploratory and with caution.

Details will be described in the statistical epidemiological analysis plan (SAP).

No formal hypothesis testing will be performed since this is a self-controlled study.

All patients who have received at least one dose of Spiolto<sup>®</sup> Respimat<sup>®</sup> will be included in the analysis; this is the treated set. All analyses will be performed on the treated set (astreated analysis). If patients have missing values for an outcome, those patients will be excluded for that outcome's analysis.

The assessment will be carried out using  $SAS^{\circledR}$  software, 9.4 version or later. The statistical characteristics presented in the end-of-text tables will be N / mean / SD / min / median / max

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

for continuous variables. Tabulations of relative and absolute frequencies will be presented for categorical variables. Incidence rates and 95% CI will be given when appropriate.

The analyses will relate to the following data as recorded in the eCRF:

- Patient demographics (age, gender, height, and weight);
- Comorbidities;
- COPD related and other concomitant medication
- History of smoking
- Reported exacerbations
- Breathlessness based on mMRC score at visit 1
- Physical Functioning based on PF-10 scores (therapeutic success at visit 2); primary outcome
- Changes from visit 1 to visit 2 in the PF-10 score; secondary outcome
- Patient satisfaction with Spiolto® Respimat® at visit 2 only; secondary outcome
- General condition of the patient: evaluated by the physician (Physician's Global Evaluation (PGE)); secondary outcome
- Adverse Drug Reactions (ADR & SADR), fatal AEs, pregnancies
- GOLD spirometric classification (1,2, 3, 4)
- GOLD patient groups (A, B, C, D)
- Details of treatment with inhaled respiratory agents before the study
- Details of treatment with respiratory agents during the study
- Reasons for ending treatment during the observation period
- Details of treatment continuation / discontinuation

For the primary outcome, the proportion of patients with therapeutic success will be presented together with the 95% confidence interval.

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The safety data will be reported according to local requirements. Statistical analysis and reporting of AEs will be descriptive in nature. Occurrences of AEs will be analyzed relative to the number of patients treated. The following parameters will be included in the safety analyses:

- Adverse events (AEs) and serious adverse events (SAEs)
- Adverse drug reactions (ADRs), serious and non-serious

If less than half of the PF-10 questions are missing for a patient, the missing values will be replaced with the mean of the other values and the PF-10 score will be calculated. If half or more than half of the PF-10 questions are missing, no score will be calculated and the PF-10 score will be marked as missing. No other missing data will be imputed. Every effort will be made to collect complete data at the specified time points. Any removal from the analysis will be documented, stating the site and patient number as well as the reason for removal.

#### 9.8 **OUALITY CONTROL**

To improve and secure data quality, automatic data checks upon data entry will be done within the eCRF. In the eCRF, plausible ranges of values for numeric data entries as well as logical data entries and listings will be provided for each entry field. Based on this, checks on completeness and plausibility will be performed upon data entry in the eCRF.

Validity of data entry thus is ensured by integrated validation checks performed by the system, indicating missing or implausible entries to the document list or investigator. All corrections will be visible from the systems audit trail.

No regular source data verification is planned in this study. However, in case of decreasing compliance (i.e. of missing data, data discrepancies, protocol violations, etc.) a for-cause audit or risk-based monitoring visit will be performed.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

The intention of this NIS is to collect new data on the physical functioning and exercise capacity of COPD patients on treatment with Spiolto<sup>®</sup> Respirat<sup>®</sup> in a real world setting.

A NIS is the most suitable instrument for obtaining information about the use of medicines in everyday therapeutic practice and thus for investigating prospectively questions in everyday therapeutic practice.

Consecutive enrolment will be employed to minimize selection bias. The entry criteria are non-restrictive which will permit the enrolment of a broad patient population. The choice of treatment is at the discretion of the investigator.

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

There are a number of different types of bias that could influence the data collection and analysis, such as selection, information, and channeling bias.

Selection bias could occur at the site level and the patient level. To minimize the site level selection bias, the goal is to have participating centers that have access to all available treatment options which are approved for use in that country for the targeted COPD patients. To minimize selection bias at the patient level, consecutive enrolment is performed. Information bias will be minimized by the use of standard eCRF, questionnaire and physicians' training on the study protocol.

An additional limitation is that the physical functioning questionnaire (PF-10) is only assessing 10 items of the full 36-Item Short Form Health Survey (SF-36).

The 7-item satisfaction scale, which is to be completed by the patient in order to measure satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup> use, is a self-designed Boehringer-Ingelheim scale, without a public source or validation status.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

#### 9.10.2 Study records

Case Report Forms (CRFs) for individual patients will be provided by the sponsor via remote data capture. All of the clinical data and site/investigator characteristics will be captured via a web-based Electronic Data Capturing system. The site staff will enter and edit the data via a secure network, with secure access features (username, password and secure identification – an electronic password system). A complete electronic audit trail will be maintained. Patients must not be identified on the eCRF by name. Appropriately coded identification (i.e. Patient numbers) must be used. All patient questionnaires will be paper-based and will be left at the site upon completion by the patient.

#### 9.10.2.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study; also current medical records must be available.

For the eCRF, the following data must be derived from source documents:

- Patient demographics (age, gender, height, and weight);
- History of smoking

# **Non-interventional Study Protocol**

#### BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Reported exacerbations
- Past COPD therapies (6 months before visit 1)
- Respirat® training (Yes/No)
- GOLD spirometric classification (1,2, 3, 4)
- GOLD patient groups (A, B, C, D)
- Concomitant diseases / Comorbidities
- Concomitant COPD and other relevant medication
- Breathlessness based on mMRC score
- Physical Functioning (PF-10) Questionnaire
- Patient Satisfaction Questionnaire
- Adverse Drug Reactions (ADR & SADR), fatal AEs, pregnancies
- Rational for Spiolto<sup>®</sup> Respimat<sup>®</sup> treatment discontinuation (if applicable)
- Details of treatment continuation / discontinuation

#### 9.10.2.2 Direct access to source data and documents

The investigator / institution will permit study-related monitoring, audits, IEC review and regulatory inspection, providing direct access to all related source data / documents. eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities (e.g. AEMPS). The Clinical Research Associate (CRA) / on site monitor and auditor may review all eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in section 9.10.2.1

### 9.10.3 Completion of study

The EC/competent authority will be notified about the end of the study (last patient out) or early termination of the study.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, and as close as possible to the standards of the International Conference of Harmonisation (ICH) Tripartite Guideline for Good Clinical Practice (GCP), Guidelines for Good Epidemiological Practice (GEP) [R10-4560], Good Pharmacoepidemiology Practice (GPP) [R09-0182], relevant BI Standard Operating Procedures (SOPs) and local regulation applicable for observational studies "Orden SAS/3470/2009de 16 de diciembre, por la que se publican las directrices sobre estudios postautorización de tipo observacional para medicamentos de uso humano".

Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol.

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

Insurance Cover: as non-interventional study and according the local regulations the insurance policy is not applicable.

#### 10.1 Study approval, patient information and informed consent

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments. According local regulation, annual follow up reports will be send to competent authorities.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative). Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorized monitors (CML/CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IEC members, and by inspectors from regulatory authorities.

### **Boehringer Ingelheim**

Page 26 of 41

# Non-interventional Study Protocol BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.2 Statement of confidentiality

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IEC and the regulatory authorities, i.e. the competent authority (CA).

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS & ADVERSE DRUG REACTIONS

#### 11.1 Definitions of adverse events

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Adverse drug reaction

An adverse drug reaction (ADR) is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse drug reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

#### Serious adverse event

A serious adverse event is defined as any AE which

- results in death,
- is life-threatening,
- requires in-patient hospitalization, or
- prolongation of existing hospitalization,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly/birth defect

Life-threatening in this context refers to a reaction in which the patient was at risk of death at the time of the reaction; it does not refer to a reaction that hypothetically might have caused death if more severe.

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be immediately life threatening or result in death or hospitalization but might jeopardize the patient or might require intervention to prevent one of the other outcomes listed above.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Adverse Event of Special Interest (AESI)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this study, e.g. the potential for AEs based on knowledge from other compounds in the same class.

No AESIs have been defined for this study.

#### 11.2 Adverse event and serious adverse event collection and reporting

The investigator shall maintain and keep detailed records of all AEs in their patient files.

#### Collection of AEs

The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorisation. Sufficient data from controlled interventional trials are available to support the evidence on the safety and efficacy of the studied BI drug. For this reason the following AE collection and reporting requirements have been defined.

The following must be collected by the investigator in the eCRF from signing the informed consent onwards until the end of the study:

- all ADRs (serious and non-serious),
- all AEs with fatal outcome (serious adverse events),

Note\*: For all patients on these data must be recorded on the AE pages in the eCRF. The separate NIS (S)AE form must in addition be used and forwarded to the local Pharmacovigilance fax as indicated in the form.

All ADRs, including those persisting after study completion must be followed up until they are resolved, have been sufficiently characterized, or no further information can be obtained.

The investigator carefully assesses whether an AE constitutes an ADR using the information below.

#### Causal relationship of adverse event

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterized by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest a reasonable causal relationship could be:

# Non-interventional Study Protocol

BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by **or attributed to the drug class**.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the **event is reproducible** when the drug is re-introduced
- **No medically sound alternative etiologies** that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically **drug-related and infrequent in the general population** not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is **no reasonable possibility of a causal relationship** could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days/weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

#### Intensity of adverse event

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated Moderate: Enough discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### Pregnancy:

In rare cases, pregnancy might occur in this study. Once a subject has been enrolled into the study with Spiolto<sup>®</sup> Respimat<sup>®</sup>, the investigator must report any drug exposure during pregnancy, which occurred in a female subject or in a partner to a male subject, to the Sponsor by means of Part A of the Pregnancy Monitoring Form. The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported by means of Part B of the Pregnancy Monitoring Form.

In the absence of a reportable AE, only the Pregnancy Monitoring Form must be completed, otherwise the NIS AE form is to be completed and forwarded (by fax) to the local Pharmacovigilance point of contact within respective timelines.

Expedited Reporting of ADRs / Fatal AEs and Drug Exposure During Pregnancy

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following must be reported by the investigator on the NIS (S)AE Form from signing the informed consent onwards until the end of the study:

Table 11.2:1 Reporting types and timelines

| Type of Report* | Timeline |
|---|---|
| All SADRs associated with Spiolto® Respimat® | immediately within 24 hours |
| All <b>AEs with fatal outcome</b> in patients exposed to Spiolto <sup>®</sup> Respimat <sup>®</sup> | immediately within 24 hours |
| All <b>non-serious ADRs</b> associated with Spiolto <sup>®</sup> Respimat <sup>®</sup> | 7 calendar days |
| All <b>pregnancy monitoring</b> forms associated with Spiolto <sup>®</sup> Respimat <sup>®</sup> | 7 calendar days |

The same timelines apply if follow-up information becomes available for the respective events. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax/email the NIS (S)AE form.

#### <u>Information required</u>

For each reportable adverse event, the investigator should provide the information requested on the appropriate eCRF pages and the NIS (S)AE form.

#### Reporting of related Adverse Events associated with any other BI drug

The investigator is encouraged to report all adverse events related to any BI drug other than the Spiolto® Respimat® according to the local regulatory requirements for spontaneous AE reporting at the investigator's discretion by using the locally established routes and AE report forms. The term AE includes drug exposure during pregnancy, and, regardless of whether an AE occurred or not, any abuse, off-label use, misuse, medication error, occupational exposure, lack of effect, and unexpected benefit.

#### 11.3 Reporting to Health Authorities

Adverse event reporting to regulatory agencies will be done by the Sponsor according to local and international regulatory requirements.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Results of this non-interventional study will be disclosed on encepp.eu and clinicaltrials.gov and a study specific publication plan will be developed to describe planned publications.

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13. **REFERENCES**

- 13.1 PUBLISHED REFERENCES Maltais F, Hamilton A, Marciniuk D, Hernandez P, Sciurba FC, Richter K, P05-09483 Kesten S. O'Donnell D Improvements in symptom-limited exercise performance over 8 h with once-daily tiotropium in patients with COPD. Chest 128 (3), 1168 - 1178 (2005) R09-0182 Guidelines for Good Pharmacoepidemiology Practices (GPP). Pharmacoepidemiology and Drug Safety 17, 200 - 208 (2008). R10-4560 Good Epidemiological Practice (GEP). IEA Guidelines for Proper Conduct of Epidemiological Reseach (2007). R13-3633 Troosters T1, Sciurba F, Battaglia S, Langer D, Valluri SR, Martino L, Benzo R, Andre D, Weisman I, Decramer M. Physical inactivity in patients with COPD, a controlled multi-center pilot-study. Respir Med. 2010 Jul; 104(7): 1005-11. doi: 10.1016/j.rmed.2010.01.012. Epub 2010 Feb 18 R15-5015 Claudio Tantucci, Denise Modina. Lung function decline in COPD. International Journal of COPD. 2012:7, 95-99. R15-4559 Katz P, Chen H, Omachi TA, Gregorich SE, Julian L, Cisternas M, Balmes J, Blanc PD Therole of physical inactivity in increasing disability among older adults with obstructive airway disease. J Cardiopulm Rehabil Prev 31 (3), 193 - 197 (2011) Maltais F, LeBlanc P, Simard C, Jobin J, Berube C, Bruneau J, Carrier L. R15-4561 Belleau R Skeletalmuscle adaptation to endurance training in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med 154, 442 -447 (1996) R15-4564 Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM Regularphysical activity reduces hospital admission and mortality in chronic obstructive
- pulmonary disease: a population based cohort study. Thorax 61, 772 778 (2006)
- P10-07776 Bouyssou T, Casarosa P, Naline E, Pestel S, Konetzki I, Devillier P, Schnapp A. Pharmacological characterization of olodaterol, a novel inhaled beta2adrenoceptor agonist exerting a 24-hour-long duration of action in preclinical models. J Pharmacol Exp Ther 334 (1), 53 - 62 (2010)
- P10-09337 Bouyssou T, Schnapp A, Casarosa P, Pieper MP. Addition of the new oncedaily LABA BI 1744 to tiotropium results in superior bronchoprotection in pre-clinical models. ATS 2010, 106th Int Conf of the American Thoracic

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Society (ATS), New Orleans, 14 - 19 May 2010. Am J Respir Crit Care Med 181, A4445, Abstr (2010)

- P10-14042 Maltais F, Beck E, Webster D, Maleki-Yazdi MR, Seibt JV, Arnoux A, Hamilton A. Four weeks once daily treatment with tiotropium + olodaterol (BI 1744) fixed dose combination compared with tiotropium in COPD patients. 20th Ann Cong of the European Respiratory Society (ERS), Barcelona, 18 22 Sep 2010. Eur Respir J 36 (Suppl 54), 1014S, Abstr 5557 (2010)
- P11-07720 Casarosa P, Kollak I, Kiechle T, Ostermann A, Schnapp A, Kiesling R, Pieper M, Sieger P, Gantner F. Functional and biochemical rationales for the 24-hour-long duration of action of olodaterol. J Pharmacol Exp Ther 337 (3), 600 609 (2011)
- P13-02357 Aalbers R, Maleki-Yazdi MR, Hamilton A, Waitere-Wijker S, Pivovarova A, Schmidt O, Bjermer L. Dose-finding study for tiotropium and olodaterol when administered in combination via the Respirat inhaler in patients with COPD. 22nd Ann Cong of the European Respiratory Society (ERS), Vienna, 1 5 Sep 2012. Eur Respir J 40 (Suppl 56), 525S 526S, Abstr P2882 (2012)
- P13-04267 Cooper CB, Celli BR, Jardim JR, Wise RA, Legg D, Guo J, Kesten S. Treadmill endurance during 2-year treatment with tiotropium in patients with COPD: a randomized trial. Chest 144 (2), 490 497 (2013)
- P13-05794 Tashkin DP, Ferguson GT. Combination bronchodilator therapy in the management of chronic obstructive pulmonary disease. Respir Res (Lond) 14, 49 (2013)
- P13-11341 Koch A, Paggiaro P, Hamilton A, Hart L, Korducki L, Salvo MC de, Pizzichini E. Symptomatic benefit of olodaterol QD delivered via Respimat vs placebo and formoterol BID in patients with COPD: combined analysis from two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11345 Koch A, Pizzichini E, Hamilton A, Hart L, Korducki L, Salvo MC de, Paggiaro P. Lung function efficacy of olodaterol QD delivered via Respirat vs placebo and formoterol BID in patients with COPD: two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11346 Ferguson G, Feldman G, Hofbauer P, Hamilton A, Allen L, Korducki L, Sachs P. Lung function efficacy of olodaterol QD delivered via Respirat in COPD patients: results from two 48-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 11 Sep 2013
- P13-11467 Lange P, Aumann JL, Derom E, Hamilton A, Tetzlaff K, Ting N, Noord JA van. The 24-h FEV1 time profile of olodaterol QD delivered via Respirat in

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

COPD: results from two 6-week studies. 23rd Ann Cong of the European Respiratory Society (ERS), Barcelona, 7 - 11 Sep 2013

- P13-14109 Maltais F, Kirsten AM, Hamilton A, Sousa D de, Wang F, Decramer M. Evaluation of the effects of olodaterol on exercise endurance in patients with COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 31 Oct 2013. Chest 144 (4) (Suppl), 748A, Abstr (2013)
- P13-14112 Feldman G, Bernstein JA, Hamilton A, Nivens C, LaForce C. The 24-hour FEV1 time profile of olodaterol once daily (QD) via Respimat and formoterol twice daily (BID) via Aerolizer in patients with COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 31 Oct 2013. Chest 144 (4) (Suppl), 749A, Abstr (2013)
- P14-01052 Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (updated 2014). http://www.goldcopd.org/uploads/users/files/GOLD\_Report\_2014.pdf (access date: 22 January 2014); Global Initiative for Chronic Obstructive Lung Disease (GOLD) (2014)
- P14-12073 Bouyssou T, Casarosa P, Pieper M, Schnapp A, Gantner F. Synergistic bronchoprotective activity of the long-acting beta 2-agonist olodaterol with tiotropium (long-acting M3 antagonist) and ciclesonide (inhaled steroid) on the ovalbumin-induced bronchoconstriction in anaesthetized guinea pigs. ERJ September 1, 2011 vol. 38 no. Suppl 55 3451
- P13-14109 Maltais F, Kirsten AM, Hamilton A, Sousa D de, Wang F, Decramer M Evaluation of the effects of olodaterol on exercise endurance in patients with COPD: results from two 6-week studies. Chest 2013, 79th Ann Mtg of the American College of Chest Physicians, Chicago, 26 31 Oct 2013 Chest 144 (4) (Suppl), 748A, Abstr (2013)
- P15-03349 Buhl R, Maltais F, Abrahams R, Bjermer L, Derom E, Ferguson G, Flezar M, Hébert J, McGarvey L, Pizzichini E, Reid J, Veale A, Grönke L, Hamilton A, Korducki L, Tetzlaff K, Waitere-Wijker S, Watz H, Bateman E. Tiotropium and olodaterol fixed-dose combination versus mono-components in COPD (GOLD 2–4) Eur Respir J 2015; DOI: 10.1183/09031936.00136014
- P15-04531 Kai-Bichael Beeh, et al. The 24-h lung-function profile of once-daily tiotropium and olodaterol fixed-dose combination in chronic obstructive pulmonary disease. Elsevier Ltd, 2015. 1094-5539
- P94-1346 Bone R, et al. In chronic obstructive pulmonary disease, a combination of ipratropium and albuterol is more effective than either agent alone: an 85-day multicenter trial. Chest 105 (5), 1411 1419 (1994)

# **Boehringer Ingelheim**

## Page 35 of 41

# Non-interventional Study Protocol BI Study Number 1237.58

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13.2 UNPUBLISHED REFERENCES

Not applicable

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

The stand-alone documents for this non-interventional study are:

- Informed Consent Form
- PF-10 Questionnaire based on SF-36
- Breathlessness Scale (mMRC)
- Patient Satisfaction Survey
- Statistical Analysis Plan (SAP)
- Data Management Plan (DMP)
- Serious Adverse Event Report in Non-Interventional Studies (NIS (S)AE Form)
- Pregnancy Monitoring Form
- Publication Plan

All of the above documents will be archived in the Trial Master File in its original master version.

c10705101-01

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ANNEX 3. ADDITIONAL INFORMATION**

1. Physical Functioning Questionnaire (PF-10) based on the 36-Item Short Form Survey.

The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not limited at all |
|---|---|---|---|---|
| a | <u>Vigorous activities</u> , such as running, lifting heavy objects, participating in strenuous sports | 1 | 2 | 3 |
| b | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 |
| С | Lifting or carrying groceries | 1 | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| e | Climbing one flight of stairs | 1 | 2 | 3 |
| f | Bending, kneeling, or stooping | i | 2 | 3 |
| g | Walking more than a mile | 1 | 2 | 3 |
| h | Walking several hundred yards | 1 | 2 | 3 |
| i | Walking one hundred yards | 1 | 2 | 3 |
| j | Bathing or dressing yourself | 1 | 2 | 3 |

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. <u>Modified Medical Research Council (mMRC) Questionnaire for Assessing the Severity of Breathlessness (\*)</u>

Please circle the number which best describes your grade of breathlessness.

| I only get breathless with strenuous exercise. | 0 |
|---|---|
| I get short of breath when hurrying on the level or walking up a slight hill. | 1 |
| I walk slower than people of the same age on the level because of breathlessness, or have to stop for breath when walking at my own pace on the level. | 2 |
| I stop for breath after walking about 100 meters or after a few minutes on level. | 3 |
| I am too breathless to leave the house or I am breathless when dressing or undressing. | 4 |

(\*) Bestall J.C. et al. Thorax. 1999 Jul;54(7):581-6. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease.

From the *Global Strategy for the Diagnosis, Management and Prevention of COPD*, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2016. Available from: <a href="http://www.goldcopd.org/">http://www.goldcopd.org/</a>. (accessed on March 2016).

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. Patient Satisfaction Questionnaire

| Please choos | se the number | which best d | escribes your | satisfaction v | with Spiolto® | Respimat <sup>®</sup> . |
|---|---|---|---|---|---|---|
| What is you | r <u>overall satis</u> | sfaction with t | the Spiolto® R | despimat <sup>®</sup> tre | atment? | |
| 1 very unsatisfied | 2<br>unsatisfied | 3 rather unsatisfied | 4 neither satisfied nor unsatisfied | 5 rather satisfied | 6<br>satisfied | 7 very satisfied |
| How satisfie | d are you wit | h <u>inhaling</u> fro | om the Respin | nat <sup>®</sup> device? | | |
| 1 very unsatisfied | 2<br>unsatisfied | 3 rather unsatisfied | 4 neither satisfied nor unsatisfied | 5 rather satisfied | 6<br>satisfied | 7 very satisfied |
| How satisfie | d are you wit | h the <u>handlin</u> | g of the Respi | imat <sup>®</sup> inhalat | ion device? | |
| 1 very unsatisfied | 2<br>unsatisfied | 3 rather unsatisfied | 4 neither satisfied nor unsatisfied | 5 rather satisfied | 6<br>satisfied | 7 very satisfied |

Poor

# Non-interventional Study Protocol

BI Study Number 1237.58

c10705101-01

Excellent

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. Physicians' Global Evaluation (PGE) to be used directly within the eCRF

| General condition of the patient at the initial examination (Visit 1) |
|-----------------------------------------------------------------------|
| Please mark with a cross as applicable |

Satisfactory

| Poor | Satisfactory | Good | Excellent |
|---|---|---|---|
| 1 2 | 3 4 | 5 6 | 7 8 |
| General condition of | f the patient after approxi | imately 6 weeks of tr | eatment (Visit 2) |
| Please mark with a c | cross as applicable | | |

Good



#### APPROVAL / SIGNATURE PAGE

Document Number: c10705101 Technical Version Number: 1.0

**Document Name:** clinical-trial-protocol-version-1.0

**Title:** Assessment of physical functioning and handling of Spiolto® Respimat® in patients with chronic obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine clinical practice.

### **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval- Safety Evaluation<br>Therapeutic Area | | 13 Jun 2016 15:40 CEST |
| Approval-Medical | | 13 Jun 2016 16:13 CEST |
| Approval-Team Member Medicine | | 13 Jun 2016 16:27 CEST |
| Approval-Clinical | | 20 Jun 2016 12:01 CEST |
| Author-Trial Statistician | | 20 Jun 2016 15:29 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c10705101Technical Version Number:1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|